CLINICAL TRIAL: NCT03811717
Title: Impact of Exercise-induced Energetic Stress During an 8-hour Fast on Metabolic Regulation in Resting Human Skeletal Muscle
Brief Title: Fasting and Exercise-induced Changes in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: University of Waterloo (Other)
Responsible Party: Principal Investigator, Brendon Gurd, Associate Professor, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: QMPL_HI-01-19
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Skeletal Muscle Energetics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation concealment, assessor blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST+EX - FAST (Experimental): FAST+EX then FAST alone
  Interventions: Other: FAST+EX; Other: FAST
- FAST - FAST+EX (Experimental): FAST alone then FAST+EX
  Interventions: Other: FAST+EX; Other: FAST

INTERVENTIONS:
Other: FAST+EX — Participants will perform 2-hours of low-intensity arm exercise (8 x 15 min bouts of arm ergometer exercise separated by 10 min of rest) during an 8-hour fast.
Other: FAST — Participants will complete an 8-hour fast.

SUMMARY:
This study examines the impact of increasing energetic stress during an 8-hour fast on metabolic pathways in human skeletal muscle. Specifically, participants will undergo two 8-hour fasting sessions in a randomized crossover fashion, with the addition of low-intensity arm exercise in one of the sessions. Changes in metabolic pathways will be examined in resting (leg) muscle before, during, and after the fast.

ELIGIBILITY:
Inclusion Criteria:

* recreationally active (no more than 3 hours of weekly physical activity)
* not currently involved in a systematic training program
* body mass index < 30 kg/m2

Exclusion Criteria:

* presence of cardiometabolic disease
* taking regular oral medication
* current smoker

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Peroxisome proliferator activated receptor gamma co-activator 1-alpha (PGC-1α) messenger ribonucleic acid (mRNA) expression | 15 min before fast; after 4 and 8 hours of fasting
  PGC-1α gene expression (indirect indicator of PGC-1α activity)

SECONDARY OUTCOMES:
Catecholamine concentrations | 15 min before fast; after exercise; after 4 and 8 hours of fasting
  Epinephrine and norepinephrine concentrations in plasma samples
Glucose and insulin concentrations | 15 min before fast; after 4 and 8 hours of fasting
  Glucose and insulin concentrations in plasma samples
total and phosphorylated AMP activated protein kinase (AMPK) | 15 min before fast; after 4 and 8 hours of fasting
  active AMPK relative to total AMPK protein content
total and phosphorylated SIRT-1 | 15 min before fast; after 4 and 8 hours of fasting
  active SIRT-1 relative to total SIRT1 protein content
total and phosphorylated mammalian target of rapamycin (mTOR) | 15 min before fast; after 4 and 8 hours of fasting
  active mTOR relative to total mTOR protein content
total and phosphorylated Akt/Protein Kinase B | 15 min before fast; after 4 and 8 hours of fasting
  active Akt relative to total Akt protein content
total and phosphorylated acetyl coenzyme A carboxylase (ACC) | 15 min before fast; after 4 and 8 hours of fasting
  active ACC relative to total ACC protein
total and phosphorylated p38 mitogen activated protein kinase (MAPK) | 15 min before fast; after 4 and 8 hours of fasting
  active p38 MAPK relative to total p38 MAPK protein
phosphorylated protein kinase A (PKA) substrates | 15 min before fast; after 4 and 8 hours of fasting
  phosphorylated PKA substrates (indirect measure of PKA activity)
acetylated p53 | 15 min before fast; after 4 and 8 hours of fasting
  p53 acetylation status (indirect measure of SIRT-1 deacetylase activity)
Sirtuin 1 (SIRT1) mRNA expression | 15 min before fast; after 4 and 8 hours of fasting
  gene expression of the deacetylase enzyme SIRT1
Sirtuin 3 (SIRT3) mRNA expression | 15 min before fast; after 4 and 8 hours of fasting
  gene expression of the deacetylase enzyme SIRT3
Pyruvate dehydrogenase kinase isoenzyme 4 (PDK4) mRNA expression | 15 min before fast; after 4 and 8 hours of fasting
  gene expression of the PGC-1α target PDK4
p53 mRNA expression | 15 min before fast; after 4 and 8 hours of fasting
  gene expression of the tumour suppressor protein p53
Leucine rich pentatricopeptide repeat containing protein (LRP130) mRNA expression | 15 min before fast; after 4 and 8 hours of fasting
  gene expression of RNA-binding protein LRP130
General control non-repressible 5 (GCN5) mRNA expression | 15 min before fast; after 4 and 8 hours of fasting
  gene expression of the acetyltransferase GCN5
PGC-1α protein content | 15 min before fast; after 4 and 8 hours of fasting
  Protein content of the transcriptional co-activator PGC-1α
Cytochrome C oxidase subunit 4 (COX-IV) protein content | 15 min before fast; after 4 and 8 hours of fasting
  Protein content of the mitochondrial enzyme COX subunit 4
Intramuscular glycogen content | 15 min before fast; after 4 and 8 hours of fasting
  Muscle glycogen content
Intramuscular triglyceride (IMTG) content | 15 min before fast; after 4 and 8 hours of fasting
  Muscle IMTG content

CONTACTS AND LOCATIONS:
Overall Officials: Brendon J. Gurd, PhD, Principal Investigator — Queen's University
Locations (1):
- School of Kinesiology and Health Studies, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No